CLINICAL TRIAL: NCT04125706
Title: Locally Delivered Antibiotics for the Treatment of Periodontitis Topical Doxycycline Versus Minocycline Gels as an Adjunct to Mechanical Treatment
Brief Title: Locally Delivered Antibiotics for the Treatment of Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Sasha Suliman, lecturer, Riyadh Elm University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRP/2019/53
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Two parallel groups will receive two different locally delivered antibiotics
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mincycline hydrochloride 2% oral gel (Experimental): Minocycline will be delivered locally in the periodontal pocket.
  Interventions: Drug: Minocycline Topical
- Metronidazole hylcate 0.75 % oral gel (Experimental): Metronidazole gel will be delivered locally in the periodontal pocket.
  Interventions: Drug: Metronidazole Topical Gel

INTERVENTIONS:
Drug: Minocycline Topical — Minocycline will be delivered locally in the periodontal pocket
  Other Names: Dentomycin oral gel will be delivered locally in the periodontal pocket
  Arms: Mincycline hydrochloride 2% oral gel
Drug: Metronidazole Topical Gel — Metronidazole will be delivered locally in the periodontal pocket
  Other Names: Roza 0.75% will be delivered locally in the periodontal pocket
  Arms: Metronidazole hylcate 0.75 % oral gel

SUMMARY:
The sample consists of patients with moderate to severe periodontitis who will be subjected to machanical therapy in combination to local antibiotics. The participants will be divided into two groups, mechanical therapy with metronidazole hyclate, and mechanical therapy with minocycline hydrochloride. Both antibiotics will be delivered locally as gels. Outcome measures include probing pocket depth and several gingival indices. IL6 will be also measured for all participants.

DETAILED DESCRIPTION:
Forty-four patients in the age group of 25-50 years (males and females) who are suffering from periodontitis with almost similar probing depth bilaterally (≥ 6 mm) at the selected sites and exhibiting bleeding on probing.

A written informed consent will be taken from the patients prior to the study.

Each patient will be recalled 4 weeks after completion of both sides supra-gingival scaling, which formed the baseline visit. Plaque scores will be brought to zero, and the probing pocket depth and gingival index, will be recorded on the proforma specially prepared for the purpose.

The selected treatment sites will be then divided into two groups, and sub-gingival SRP will be performed prior to the delivery of the drugs at the test sites.

* Group I: Consist of periodontal pockets on the left side of maxillary or mandibular arch and received sub-gingival Minocycline 2% gel.
* Group II: Consist of periodontal pockets on the left side of maxillary or mandibular arch and received Metronidazole 0.75% gel.

The right side will be left as a control in both groups Patients will be recalled after 6 weeks from the baseline visit to record the plaque index, gingival index, bleeding index and probing depth (UNC probe 12 mm).

Statistical Analysis:

The unit of measurement in this study is the site, rather than the subject. Student-t test was To compare between Group 1 (Minocycline 2 %) and Group 2 (Metronidazole 0.75 %), Data will check for normality, if the data normally distributed Independent t-test will use to test if there any significant differences between groups, otherwise if not normally Mann -Whitney U-test (Non-parametric) will use to detects the difference.

To achieve 80% power of statistical test to detect the differences between Metronidazole and Minocycline With 5 % level of significant, 19.6 reduction in probing depth (previous study-vi) and standard deviation of 0.23, using the following formula.

n=(2σ^2 〖(Z_(β+Z_(1-α/2) ))〗^2)/d^2 22 per group (minimum sample size) where: σ =0.23 Zβ =0.84 Z(1-α/2) =1.96, d= 19.6%

For objective 2, the statistical test in case of normal data distribution will be paired t test or will use Willcoxon Sign Ranked test if it not normally distributed.

To achieve 80% power of statistical test to detect the differences between Metronidazole and Minocycline. With 5% level of significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from chronic periodontitis with almost similar probing depth bilaterally (≥
* 6 mm) at the selected sites and exhibiting bleeding on probing Patients with no caries and restorations on the selected teeth
* Patients showing effective individual oral hygiene.

Exclusion Criteria:

Patients presenting with history of intake of local and/or systemic antibiotic therapy for the last 3 months

* Patients with known systemic and debilitating diseases (Muscular Dystrophy)
* Patients presenting with known adverse reactions to any component of the test agent
* Patients on anticoagulant therapy
* Pregnant and lactating females
* Smokers
* Patients in a regular use of mouth wash

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
plaque index | Baseline to six weeks
  To measure the state of oral hygiene as:
  0 = No plaque in the gingival area
  1. = A film of plaque adhering to the free gingival margin and adjacent of the tooth
  2. = Moderate accumulation of soft deposits within the gingival pocket
  3. = Abundance of soft matter within the gingival pocket
  The Plaque Index is the four gingival areas of the tooth (buccal, lingual/palatal, mesial, distal) given a score from 0-3 and scores were added and divided by four. The plaque index for the individual was obtained by adding the indices for the teeth and divide by the number of teeth examined.
gingival index | Baseline to six weeks
  To assess the gingival condition and record qualitative chances in the gingiva as:
  0 = Normal gingiva
  1. = Mild inflammation - slight change in color and slight edema but no bleeding on probing.
  2. = Moderate inflammation - redness, edema and glazing, bleeding on probing
  3. = Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.
  The bleeding will be assessed by gently probing along the wall of the soft tissue of the gingival sulcus. To get the gingival index for the tooth, the four areas of the tooth (buccal, lingual/palatal, mesial, distal) are scored by the sum and divided by four. The gingival index for the individual will be obtained by adding the indices of the teeth and divided by the number of teeth examined.
probing depth | Baseline to six weeks
  The distance from the gingival margin to base of the sulcus. Will be measured at six sites per tooth (mesio-buccal, buccal, disto-buccal, disto-lingual, lingual and mesio-lingual) at all teeth with UNC-15 probe.
IL6 | Baseline to six weeks
  In healthy subjects it ranges from 0.5-5 pg/ml In eosinophilic subjects it ranges from 3-18pg/ml in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Sasha M Suliman, MSc, Principal Investigator — Ar Riyad, Saudi Arabia, 11681

IPD SHARING:
Plan to Share IPD: No